CLINICAL TRIAL: NCT02212522
Title: Genetic and Environmental Risk Factors of Type 1 Autoimmune Diabetes and Its Early Complications. French Multicentric Cohort of Diabetic Patients.
Brief Title: Genetic and Environmental Risk Factors of Type 1 Autoimmune Diabetes and Its Early Complications
Acronym: ISIS-DIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de Génotypage (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOM 08049
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus; Insulin-Dependent
Keywords: Diabetes Mellitus; Insulin-Dependent; Genome-Wide Association Study; Environment-Wide Association Study; Predisposition; Complications
MeSH Terms: conditions — Diabetes Mellitus; Disease Susceptibility | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Isis-Diab patients: French T1D patients with genetic data (GWAS), and environmental data (questionnaire and environmental databases), clinical data
  Interventions: Other: Collect of environmental data on T1D patients before diagnosis; Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS); Other: Collect of clinical data on the disease and its evolution
- Isis-Diab controls: French control population with genetic data (GWAS) and environmental data (questionnaire and environmental databases
  Interventions: Other: Collect of environmental data on French controls (age-matched for T1D patients); Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS)

INTERVENTIONS:
Other: Collect of environmental data on T1D patients before diagnosis — Questionnaires on large environment during mother's pregnancy and patient's childhood, health book copies, addresses' geolocation, quantification of viral exposures using Sentinel Network data
  Groups: Isis-Diab patients
Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS) — Collect of blood samples for DNA extraction and genetic characterization (GWAS) on Illumina platform (Centre National de Genotype)
  Groups: Isis-Diab patients
Other: Collect of clinical data on the disease and its evolution — Collect of clinical data on the disease and its evolution every 6 months after enrollment
  Groups: Isis-Diab patients
Other: Collect of environmental data on French controls (age-matched for T1D patients) — Questionnaires on large environment during mother's pregnancy and patient's childhood, health book copies, addresses' geolocation, quantification of viral exposures using Sentinel Network data
  Groups: Isis-Diab controls
Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS) — Collect of blood samples for DNA extraction and genetic characterization (GWAS) on Illumina platform (Centre National de Genotype)
  Groups: Isis-Diab controls

SUMMARY:
The aim of this study is to complete the identification of genetic factors (G) and to undertake the search of environmental factors (E) predisposing to type 1 diabetes (T1D) by constituting a cohort of 3500 T1D patients and a control cohort. We will use the base of G analysis (whole genome genotyping done once a patient using methods conually updated at Centre National de Genotype) and innovative E analysis to develop the following long term objectives :

* Identify G and E factors influencing the process of remaining beta cells' destruction during the first 3 years after diagnosis (subgroup of T1D patients with a 0-3 years diabetes duration);
* Identify G factors (pharmacogenomics) of the individual response to insulin using the effective insulin dose as a phenotype over a period of 2 years (subgroup of T1D patients with negative C-peptide and well managed diabetes);
* Undertake a prospective research of G and E risk factors of "death in bed" syndrome in diabetic adolescents;
* Undertake a prospective research of G and E risk factors of incipient glomerular microangiopathy (regule measurement of microalbuminuria).

DETAILED DESCRIPTION:
Still recognized in youth only at a stage of complete beta-cell mass destruction and insulin deficiency, autoimmune T1D remains a source of major morbidity through daily life and chronic angiopathic complications despite a better glycemic control. T1D onset is now predominantly pediatric, since its incidence shows a rapid and continuous increase in young European children, due to unknown emerging environmental changes, creating a major need for discoveries in the environmental field. Finding avoidable E factors can allow T1D prevention in the whole children population. Lack of infectious exposures ("the hygiene hypothesis"), viruses, early nutrition, or other factors have been suspected, but E causes of T1D remain a black box, as for most human diseases, that should now be approached more systematically and with respect to gene-environment interactions.

The aim of our study is to complete the identification of genetic factors (G) and to undertake the search of environmental factors (E) predisposing to type 1 diabetes (T1D) by constituting a cohort of 3500 T1D patients and a control cohort. We will use the base of G analysis (whole genome genotyping done once a patient using methods conually updated at Centre National de Genotype) and innovative E analysis to develop the following long term objectives :

* Identify G and E factors influencing the process of remaining beta cells' destruction during the first 3 years after diagnosis (subgroup of T1D patients with a 0-3 years diabetes duration);
* Identify G factors (pharmacogenomics) of the individual response to insulin using the effective insulin dose as a phenotype over a period of 2 years (subgroup of T1D patients with negative C-peptide and well managed diabetes);
* Undertake a prospective research of G and E risk factors of "death in bed" syndrome in diabetic adolescents;
* Undertake a prospective research of G and E risk factors of incipient glomerular microangiopathy (regule measurement of microalbuminuria).

We propose to constitute a French multicentric cohort of T1D patients, well phenotyped by 3 data types : genetic, environmental and clinical data. The data collection scheme includes at entry a comprehensive 850 items environmental questionnaire for all subjects and a full genotyping with at least 500,000 SNPs until whole-genome sequencing can be deployed by CNG-CEA. Every 6 months, a standardized clinical assessment is made in patients (a WEB application ensuring this standardization has already been developed). Personal address(es) will be collected and geocoded, then mapped with environmental geographic information systems (GIS).

With environmental modelling, the high dimensionality analyses (HDA) constitutes one of the main originality of ISIS-DIAB approaches of translational research. HDA will face not only a massive mass of data, but data of a remarkable diversity (genomic variants, environmental items from questionnaires, environmental data bases mapped to patient address, space-time items, characteristics of social environment, clinical phenotypes etc). A given genotype (defined by many genomic variants) will predispose to T1D only in a given environmental context (defined possibly by a number of factors) and induce a given type of autoimmune process (age of onset, rate of destruction, biomarkers). Since T1D is both multifactorial and heterogeneous, causal factors may interact in a considerable number of scenarii, thus platforms which study these factors should obviously interact. Without HDA, each platform would be left faced with its own data. The chef d'orchestre has to be HDA, to integrate the massive amounts of data and draw networks of causality. Technological advances in HDA developed in other fields of sciences, business and economics (forecasting technology) will be transferred to biomedical research through ISIS-DIAB. French have a strong tradition of high-level maths in this area. We designed the ISIS-DIAB cohort and collection of data to feed HDA with multidisciplinary data. In ISIS-DIAB program, HDA will identify the variables that have the most predictive value on several outcomes (not confined to T1D causality).

ELIGIBILITY:
Inclusion Criteria:

* Insulin-dependent diabetes
* Patients older than 6 months at inclusion
* European or North African geographical origin (defined by the birthplaces of the 4 grandparents), for the purpose of genetic homogeneity of the cohort
* Anti-GAD, IA2, and insulin autoantibodies, that are present only in the first year of the disease evolution, are not a criterion of absolute inclusion (low risk of error) but will be noted if they were searched at diagnosis
* Informed consent dated and voluntarily signed (patient and/or parents)

Exclusion Criteria:

* Non-insulin dependent diabetes
* MODY
* Severe psychological problems, co-morbidities that could possibly invalidate informed consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients: T1D patients are enrolled into the Isis-Diab cohort, continuously, from 110 clinical diabetes centers distributed over the whole France territory. Inclusion in the cohort occurs most often soon after the initial diagnosis of T1D. This diagnosis is made according to classical criteria of autoimmune T1D.
  Controls: we will recruit age-matched controls among friend patients' families and among cases admitted in the participating centers for benign transient intercurrent events.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2004-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Genetic and environmental risk factors of T1D predisposition | 10 years

SECONDARY OUTCOMES:
Genetic and environmental risk factors of T1D complications | 10 years
  Regular measurement of microalbuminuria
Identify G and E factors influencing the process of remaining beta cells' destruction during the first 3 years after diagnosis | 5 years
  Subgroup of T1D patients with a 0-3 years diabetes duration
Identify G factors (pharmacogenomics) of the individual response to insulin using the effective insulin dose as a phenotype over a period of 2 years | 4 years
  Subgroup of T1D patients with negative C-peptide and well managed diabetes
Undertake a prospective research of G and E risk factors of "death in bed" syndrome in diabetic adolescents | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUGNERES, MD-PhD, Principal Investigator — Inserm U986/ Pediatric endocrinology department of the Bicêtre hospital
Locations (1):
- Inserm U986, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balazard F, Le Fur S, Valtat S, Valleron AJ, Bougneres P; Isis-Diab collaborative group; Thevenieau D, Chatel CF, Desailloud R, Bony-Trifunovic H, Ducluzeau PH, Coutant R, Caudrelier S, Pambou A, Dubosclard E, Joubert F, Jan P, Marcoux E, Bertrand AM, Mignot B, Penformis A, Stuckens C, Piquemal R, Barat P, Rigalleau V, Stheneur C, Fournier S, Kerlan V, Metz C, Fargeot-Espaliat A, Reznic Y, Olivier F, Gueorguieva I, Monier A, Radet C, Gajdos V, Terral D, Vervel C, Bendifallah D, Signor CB, Dervaux D, Benmahammed A, Loeuille GA, Popelard F, Guillou A, Benhamou PY, Khoury J, Brossier JP, Bassil J, Clavel S, Le Luyer B, Bougneres P, Labay F, Guemas I, Weill J, Cappoen JP, Nadalon S, Lienhardt-Roussie A, Paoli A, Kerouedan C, Yollin E, Nicolino M, Simonin G, Cohen J, Atlan C, Tamboura A, Dubourg H, Pignol ML, Talon P, Jellimann S, Chaillous L, Baron S, Bortoluzzi MN, Baechler E, Salet R, Zelinsky-Gurung A, Dallavale F, Larger E, Laloi-Michelin M, Gautier JF, Guerin B, Oilleau L, Pantalone L, Lukas C, Guilhem I, De Kerdanet M, Wielickzo MC, Priou-Guesdon M, Richard O, Kurtz F, Laisney N, Ancelle D, Parlier G, Boniface C, Bockel DP, Dufillot D, Razafimahefa B, Gourdy P, Lecomte P, Pepin-Donat M, Combes-Moukhovsky ME, Zymmermann B, Raoulx M, Dumont AG. Association of environmental markers with childhood type 1 diabetes mellitus revealed by a long questionnaire on early life exposures and lifestyle in a case-control study. BMC Public Health. 2016 Sep 29;16(1):1021. doi: 10.1186/s12889-016-3690-9. PMID 27682602